CLINICAL TRIAL: NCT05482308
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, CROSSOVER, SINGLE DOSE STUDY TO ESTIMATE THE RELATIVE BIOAVAILABILITY OF VARIANT 12.2 MG TAFAMIDIS FREE ACID TABLETS AND PROPOSED COMMERCIAL 12.2 MG TAFAMIDIS FREE ACID TABLETS ADMINISTERED UNDER FASTED CONDITIONS IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Compare Two Tablet Forms of Tafamidis in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B3461102; 2022-001833-35 (EudraCT Number)
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Results first posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test tablet followed by Reference tablet (Experimental): On Day 1 of each period, participants will receive a single dose of 1 of the tafamidis formulations. Each period is separated by a washout of at least 16 days between administration of study drug.
  Interventions: Drug: Tafamidis free acid tablet (Test); Drug: Tafamidis free acid tablet (Reference)
- Reference tablet followed by Test tablet (Experimental): On Day 1 of each period, participants will receive a single dose of 1 of the tafamidis formulations. Each period is separated by a washout of at least 16 days between administration of study drug
  Interventions: Drug: Tafamidis free acid tablet (Test); Drug: Tafamidis free acid tablet (Reference)

INTERVENTIONS:
Drug: Tafamidis free acid tablet (Test) — Variant 12.2 mg tafamidis free acid tablet (Test)
Drug: Tafamidis free acid tablet (Reference) — Proposed commercial 12.2 mg tafamidis free acid tablet (Reference)

SUMMARY:
The purpose of this clinical trial is to compare the amount of tafamidis in blood after taking two different tablet forms of tafamidis

This study is seeking healthy participants over the age of 18.

All participants in the study will receive one tablet of study medicine on the first day, then receive one dose of the other tablet form 16 days later.

We will compare the amounts in blood for 8 days after taking each dose of the study medicine.

Participants will take part in this study for about 80 days. The first visit is a screening visit to ensure that participants are appropriate for the study. Up to 28 days later, they will visit the study clinic twice (and stay overnight in the clinical research center for 8 nights each time). The study team will also call participants over the phone 28 to 35 days after the last dose of medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 years or older (or the minimum age of consent in accordance with local regulations) at screening.
2. Healthy female participants of nonchildbearing potential and/or male participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, and laboratory tests.
3. Body Mass Index of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

Medical Conditions:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

   * Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
   * History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, HBcAb, or HCVAb. Hepatitis B vaccination is allowed.
   * Hypersensitivity to any component of the formulations
2. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to COVID-19 pandemic (eg, Contact with positive case, residence, or travel to an area with high incidence) that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

   Prior/Concomitant Therapy:
3. Use of prescription or nonprescription drugs, dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention. (Refer to Section 6.9 Prior and Concomitant Therapy for additional details).
4. Current use of any prohibited concomitant medication(s) or participant unwilling/unable to use a permitted concomitant medication(s). Refer to Section 6.9 Prior and Concomitant Therapy.

   Prior/Concurrent Clinical Study Experience:
5. Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).

   Diagnostic Assessments:
6. A positive urine drug test.
7. Screening seated BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of seated rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
8. Standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF >450 ms, complete LBBB, signs of an acute or indeterminate age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second or third degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the uncorrected QT interval is >450 ms, this interval should be rate-corrected using the Fridericia method only and the resulting QTcF should be used for decision making and reporting. If QTcF exceeds 450 ms, or QRS exceeds 120 ms, the ECG should be repeated twice and the average of the 3 QTcF or QRS values used to determine the participant's eligibility. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding a participant.
9. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

   * AST or ALT level ≥ 1.5 × ULN;
   * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.

   Other Exclusion Criteria:
10. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit, or 3 ounces (90 mL) of wine).
11. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
12. History of sensitivity to heparin or heparin induced thrombocytopenia.
13. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of the protocol.
14. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.
15. Use of tobacco or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3461102

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a 2-period,fixed-sequence crossover study. A total of 12 participants were randomized and assigned to study treatments.
Groups:
- Variant 12.2 mg Tafamidis Free Acid Tablet ->Proposed Commercial 12.2 mg Tafamidis Free Acid Tablet: Participants received 1 dose of Variant 12.2 mg Tafamidis free acid tablet on Day 1 of Period 1, then after a washout of at least 16 days, participants received 1 dose of Proposed commercial 12.2 mg tafamidis free acid tablet.
- Proposed Commercial 12.2 mg Tafamidis Free Acid Tablet ->Variant 12.2 mg Tafamidis Free Acid Tablet: Participants received 1 dose of Proposed commercial 12.2 mg tafamidis free acid tablet on Day 1 of Period 1 ,then after a washout of at least 16 days, participants received 1 dose of Variant 12.2 mg Tafamidis free acid tablet.
Period: Overall Study
Arm/Group | Variant 12.2 mg Tafamidis Free Acid Tablet ->Proposed Commercial 12.2 mg Tafamidis Free Acid Tablet | Proposed Commercial 12.2 mg Tafamidis Free Acid Tablet ->Variant 12.2 mg Tafamidis Free Acid Tablet
Started | 6 | 6
Completed | 5 | 5
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — No longer meets eligibility criteria | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants enrolled in the study.
Groups:
- Variant 12.2 mg Tafamidis Free Acid Tablet->Proposed Commercial 12.2 mg Tafamidis Free Acid Tablet: Participants received 1 dose of Variant 12.2 mg Tafamidis free acid tablet on Day 1 of Period 1, then after a washout of at least 16 days, participants received 1 dose of Proposed commercial 12.2 mg tafamidis free acid tablet.
- Proposed Commercial 12.2 mg Tafamidis Free Acid Tablet->Variant 12.2 mg Tafamidis Free Acid Tablet: Participants received 1 dose of Proposed commercial 12.2 mg tafamidis free acid tablet on Day 1 of Period 1 ,then after a washout of at least 16 days, participants received 1 dose of Variant 12.2 mg Tafamidis free acid tablet.
- Total: Total of all reporting groups
Arm/Group | Variant 12.2 mg Tafamidis Free Acid Tablet->Proposed Commercial 12.2 mg Tafamidis Free Acid Tablet | Proposed Commercial 12.2 mg Tafamidis Free Acid Tablet->Variant 12.2 mg Tafamidis Free Acid Tablet | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Customized [Count of Participants; unit: Participants]
  < 18 years | 0 | 0 | 0
  18-44 years | 4 | 3 | 7
  45-64 yerars | 2 | 3 | 5
  >= 65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 5 | 5 | 10
  Race: Black or African American | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of Tafamidis (Both Variant 12.2 mg Tafamidis Free Acid Tablet and Proposed Commercial 12.2 mg Tafamidis Free Acid Tablet)
Description: The AUCinf was determined by AUClast+ (Clast*/kel), where Clast* is the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis; kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Days 1 (Pre-dose,0.5,1,2,3,4,6,8,12 hours post dose),2,3,4,5,6,7 and 8 in both Periods 1 and 2.
Population: The PK parameter population was defined as all participants who received at least 1 dose of tafamidis and who had at least 1 of the PK parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour(h)*ng/mL
Groups:
- Variant 12.2 mg Tafamidis Free Acid Tablet (Test): Participants received 1 dose of Variant 12.2 mg Tafamidis free acid tablet, either in Period 1 or Period 2.
- Proposed Commercial 12.2 mg Tafamidis Free Acid Tablet (Reference): Participants received 1 dose of Proposed commercial 12.2 mg tafamidis free acid tablet, either in Period 1 or Period 2.
Arm/Group | Variant 12.2 mg Tafamidis Free Acid Tablet (Test) | Proposed Commercial 12.2 mg Tafamidis Free Acid Tablet (Reference)
Number analyzed (Participants) | 11 | 12
hour(h)*ng/mL | 58630 (21) | 57060 (25)
Statistical Analysis 1: Comparison: Variant 12.2 mg Tafamidis Free Acid Tablet (Test) vs Proposed Commercial 12.2 mg Tafamidis Free Acid Tablet (Reference); Test type: Other; Mixed effect model; Mixed effect model was fitted to obtain: 1.Adjusted mean differences 2.90% Confidence intervals(CI); Mean differences(Test-Reference) = 98.35, 90% CI 2-sided [92.92 to 104.10]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Tafamidis (Both Variant 12.2 mg Tafamidis Free Acid Tablet and Proposed Commercial 12.2 mg Tafamidis Free Acid Tablet)
Description: Cmax was observed directly from data.
Time Frame: Days 1 (Pre-dose,0.5,1,2,3,4,6,8,12 hours post dose),2,3,4,5,6,7 and 8 in both Periods 1 and 2.
Population: The PK concentration population was defined as all participants who receive dat least 1 dose of tafamidis and who had at least 1 measurable concentration of tafamidis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Variant 12.2 mg Tafamidis Free Acid Tablet (Test)): Participants received 1 dose of Variant 12.2 mg Tafamidis free acid tablet, either in Period 1 or Period 2.
Arm/Group | Variant 12.2 mg Tafamidis Free Acid Tablet (Test)) | Proposed Commercial 12.2 mg Tafamidis Free Acid Tablet (Reference)
Number analyzed (Participants) | 11 | 12
ng/mL | 875.2 (22) | 926.5 (22)
Statistical Analysis 1: Comparison: Variant 12.2 mg Tafamidis Free Acid Tablet (Test)) vs Proposed Commercial 12.2 mg Tafamidis Free Acid Tablet (Reference); Test type: Other; Mixed effect model; Mixed effect model was fitted to obtain: 1.Adjusted mean differences 2.90% Confidence intervals(CI); Mean difference (Test-Reference) = 91.58, 90% CI 2-sided [81.50 to 102.90]

ADVERSE EVENTS:
Time Frame: From informed consent through and including a minimum of 28 calendar days after last administration of study drug, up to 35 days.
Description: Both non-serious adverse events (NSAEs) and serious adverse events(SAEs) were recorded on the case report form (CRF).
Groups:
- Commercial 12.2 mg Tafamidis Free Acid Tablet (Reference): Participants received 1 dose of Proposed commercial 12.2 mg tafamidis free acid tablet, either in Period 1 or Period 2.
Arm/Group | Variant 12.2 mg Tafamidis Free Acid Tablet (Test)) | Commercial 12.2 mg Tafamidis Free Acid Tablet (Reference)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 6/11 | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Variant 12.2 mg Tafamidis Free Acid Tablet (Test)) (N=11) | Commercial 12.2 mg Tafamidis Free Acid Tablet (Reference) (N=12)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Vessel puncture site haematoma (General disorders) | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT05482308/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT05482308/SAP_001.pdf